CLINICAL TRIAL: NCT02546973
Title: ANCA - A Registry Based Study of Clinical Results and Health Related Quality of Life in Patients After Treatment for Anal Cancer
Brief Title: Quality of Life in Patients With Anal Cancer
Acronym: ANCA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Eva Angenete, M.D., Ph.D., Ass. Prof., Sahlgrenska University Hospital
Other Study IDs: ANCA
Record Dates: First submitted 2015-08-26; First posted 2015-09-11 (Estimated); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Anal Cancer
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with anal cancer: All patients with anal cancer during 2011-2013 will be asked to participate

SUMMARY:
A national study of a three year cohort consisting of all patients diagnosed with anal cancer in 2011- 2013 with data retrieval from three national registries: Cancer Registry, Patient registry and Cause of Death Registry all within the Swedish Board of Health and Welfare. All out- and inpatient visits with diagnoses, admission dates and discharge dates will be requested including.

Patient documentation from the concerned hospitals will be collected and data on the details of the treatment collected retrospectively in a standardised fashion using a clinical record form.

Comorbidity will be calculated using data from the Patient Registry using all main and co-diagnoses 2 years prior and then at least two years after treatment cessation.

Detailed questionnaires will be sent out once at 2-3 years and a second time at about 6 years after index treatment.

DETAILED DESCRIPTION:
Squamous cell carcinoma of the anus or "anal cancer" is an uncommon disease in the Western world. In Sweden approximately 100 patients are diagnosed each year. Most patients are treated by chemotherapy and radiation, but a small subgroup of non-responders and patients with recurrent disease undergo abdominoperineal excision with a permanent colostomy. In most reports of results these patients have a worse prognosis and a higher risk of local recurrence than anal cancer as a group(1, 2), possibly a result of a selection bias. Recently the results in a large Nordic cohort were presented, indicating that a further factor connected with successful outcome was that the patient was included in a treatment protocol(3).

A small number of patients with very small cancers are operated on primarily. This is especially true for anal margin tumours(4). However, for the most part patients will be primarily treated with radiotherapy, as their curative treatment.

In Sweden the treatment has been centralised for many years. The radiotherapy is normally a long course therapy with many smaller doses resulting in a high dose of radiation. There are well known complications such as skin problems and to some extent chronic radiation effects on deeper structures, which can result in functional side effects. If the treatment includes an abdominoperineal excision, the effects of a colostomy on quality of life as well as functional aspects of this surgical procedure are largely unknown in this group of patients. In our research group we have earlier studied large cohorts of patients who have undergone abdominoperineal excision for rectal cancer, and also unselected groups of patients with rectal cancer, studying both functional aspects and quality of life using detailed questionnaires (5, 6). Further we have results on quality of life from a cohort of Swedish inhabitants, representing men and women aged 30 to 90 years. The majority of the questions in these questionnaires are similar making comparisons possible.

In other studies within the SSORG network we have used the "Steineck concept" to investigate patient experiences of health, functional results and quality of life (7-11). We use specific questionnaires with detailed questions about experiences and symptoms asking about severity and duration as well as questions on socioeconomic functioning and life style factors (12, 13). Our experience is that patients are motivated to answer such questionnaires, with a compliance at 3 months >90% and at 12 months >85%.

ELIGIBILITY:
Inclusion Criteria:

* All patients registered with a diagnosis of anal cancer in either the Patient registry or the Cancer Registry during 2011 - 2013.

Exclusion Criteria:

* No informed consent received for participation in the questionnaire part of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with anal cancer diagnosed 2011-2013
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-09; Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
HRQL in patient's with anal cancer 3 years after diagnosis | 3 years
  To determine HRQL in patient's with anal cancer 3 years after diagnosis using a thorough questionnaire

SECONDARY OUTCOMES:
HRQL in patient's with anal cancer 6 years after diagnosis Functional aspects and symptoms | 6 years
  To determine HRQL in patient's with anal cancer 3 years after diagnosis using a thorough questionnaire
Comorbidity in the cohort prior to the diagnosis anal cancer | 3 years
Post-treatment morbidity in patients treated for anal cancer | 3 years
Type and number of surgical procedures in the patient population treated for anal cancer | 6 years
Accumulated length of hospital stay | 6 years
Differences in morbidity related to different treatments regimes | 3 and 6 yeras
Complete health economic analysis of resource consumption | 6 years
Mortality after anal cancer treatment | 3 and 6 years
Patient related personal factors that may affect HRQL measured by questionnaires | 3 years
Effect of complications on the patient's socioeconomic situation | 3 years
HRQL (measured by questionnaires) differences between patient groups such as age, gender and educational level | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Eva Angenete, M.D., Ph.D., Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Dept. of Surgery, Sahlgrenska University Hospital/Ostra, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No